CLINICAL TRIAL: NCT05691621
Title: A Prospective Observational Study of Galectin-3 in Septic and Non-septic Acute Kidney Injury
Brief Title: Galectin-3 in Septic and Non-septic Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fengyun Wang (Other)
Collaborators: Wuhan University (Other)
Responsible Party: Sponsor-Investigator, Fengyun Wang, Principal Investigator, First People's Hospital of Foshan
Organization: First People's Hospital of Foshan (Other)
Other Study IDs: FirstPeopleFoshan
Record Dates: First submitted 2023-01-08; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Blood or urine samples within 24 hours after ICU admission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- septic AKI: S-AKI: Septic patients with AKI
  Interventions: Drug: Standard Reagents, Whole Blood
- non-septic AKI: non-S AKI: Non-septic critically ill patients with AKI.
  Interventions: Drug: Standard Reagents, Whole Blood
- non-AKI Non-AKI: Critically ill patients without sepsis and AKI.
  Interventions: Drug: Standard Reagents, Whole Blood

INTERVENTIONS:
Drug: Standard Reagents, Whole Blood — All patients receive standard treatment, only their blood and urine samples are needed
  Other Names: Urine samples within 24 hours after ICU admission

SUMMARY:
Acute kidney injury (AKI) is a common critical condition with high morbidity and mortality. The level of circulating Galectin-3 (Gal3) largely depends on renal function, so it is elevated in patients with AKI or CKD; elevated Gal3 also aggravates the progression of CKD after the onset of AKI. The proinflammatory and profibrotic properties of Gal3 may render it to be one of the key molecules mediating AKI, CKD, and cardiorenal syndrome. In this prospective observational study, the investigators will explore the differences of Gal3 levels among septic AKI, non-septic AKI, and non-AKI patients and its correlation with prognosis, inflammation, and disease severity in the ICU.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common critical condition with high morbidity and mortality. Not only can AKI cause death in the acute phase, but also can it be associated with the development of chronic kidney disease (CKD) or the progression of CKD. Galectins are members of a lectin family widely expressed in vertebrates, among which galectin-3 (Gal3) is the most studied one. The level of circulating Gal3 largely depends on renal function, so it is elevated in patients with AKI or CKD; elevated Gal3 also aggravates the progression of CKD after the onset of AKI. The proinflammatory and profibrotic properties of Gal3 may render it to be one of the key molecules mediating AKI, CKD, and cardiorenal syndrome. However, the mechanisms of AKI differ from different etiologies, and the process and extent of levels of Gal3 may be also different, so its predictive value in prognosis may vary in different types of AKI. In critically ill patients, AKI is a common complication of sepsis, and sepsis is the most common trigger of AKI. In this prospective observational study, the investigators will explore the differences of Gal3 levels among septic AKI, non-septic AKI, and non-AKI patients and its correlation with prognosis, inflammation, and disease severity in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years old or more.
* 2. The patient himself or his agent is able to provide informed consent and provide adequate information for the endpoint assessment.
* 3. Renal function was stable before this onset, and there was no evidence of plasma creatinine rising by 0.3 mg/dL within 3 months of study entry and not receiving RRT.

Exclusion Criteria:

* 1. Age less 18 years old.
* 2. There were previous acute kidney injury, kidney transplantation, chronic kidney disease, or with a glomerular filtration rate of less than 30 mL/min, or hepatorenal syndrome, or pregnancy.
* 3. Patients with an expected survival time of less than 6 months.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis or AKI, or non-sepsis and non-AKI patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The levels of Gal3 | 2023-01~2023-08
  The levels of Gal3 in septic AKI, non-septic AKI, and non-AKI patients in the ICU

SECONDARY OUTCOMES:
Mortality | 2023-01~2023-08
  mortality at 28 days after ICU admission
Length of stay in the ICU | 2023-01~2023-08
  The days of patients in the ICU
Renal replacement therapy incidence | 2023-01~2023-08
  The incidence of RRT during the trial
Cardiovascular events incidence | 2023-01~2023-08
  The incidence of cardiovascular events during the trial
IL-6 | 2023-01~2023-08
  Interleukin-6
HMGB1 | 2023-01~2023-08
  High mobility group box 1
NGAL | 2023-01~2023-08
  Neutrophil gelatinase-associated lipid carrier protein
TIMP-2 | 2023-01~2023-08
  Tissue inhibitor of metalloproteinase 2

CONTACTS AND LOCATIONS:
Overall Officials: Fengyun Wang, Doctor, Principal Investigator — First People's Hospital of Foshan
Locations (1):
- Critical Care Department, First People's Hospital of Foshan, Foshan, China

IPD SHARING:
Plan to Share IPD: No